CLINICAL TRIAL: NCT00609752
Title: Adverse Effects of Glucocorticoid Therapy on Bone in Childhood Crohn's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: SHS International (Unknown); Children's Memorial Research Foundation (Unknown); St George's University Hospital Research Foundation (Unknown)
Responsible Party: Dr M S Murphy, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_06_266; EudraCT: 2006-000209-48; CTA: 21761/0213/001
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Children; Bone Density; Prednisolone; Liquid Diet Therapy; Quality of Life; Metabolic Bone Disease
MeSH Terms: conditions — Crohn Disease; Bone Diseases, Metabolic | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: prednisolone
- 2 (Active Comparator)
  Interventions: Dietary Supplement: Alicalm (polymeric liquid formula)

INTERVENTIONS:
Drug: prednisolone — Standard treatment regimens based on body weight will be used (approximately 2 mg per kg), with a stepwise dose reduction over a 10-14 week period.
  Arms: 1
Dietary Supplement: Alicalm (polymeric liquid formula) — Subjects will receive all of their nutritional requirements in the form of a nutritionally balanced polymeric feed, volume based on EAR for age. Duration of 5 to 8 weeks with subjects returning to a "normal" unrestricted diet by 10 weeks.
  Other Names: Alicalm (SHS International Ltd.)
  Arms: 2

SUMMARY:
This study will compare two current first-line treatments for childhood Crohn's Disease, steroids versus a liquid diet, and determine the effects of these treatments on bone health, quality of life and treatment efficacy.

DETAILED DESCRIPTION:
Crohn's Disease is a very serious inflammatory gut disorder that often first presents in childhood. Once present, the underlying condition remains for life. It usually responds well to medical treatment which brings about a disease 'remission' but is inclined to become active again at intervals (relapses). When it is active, children are very unwell with reduced energy, loss of appetite and distressing abdominal symptoms (pain, diarrhea, etc.). Active disease can be treated in two very different ways - either with a 3-month course of steroids (tablets), or with a 6-week course of so called "liquid diet therapy (LDT)." With LDT, children receive all of their nutrition in liquid form. Both treatments have advantages and disadvantages. Both are quite effective, often controlling symptoms within days. Steroids may cause various side effects including thinning of bones (osteoporosis) with increased risk of fractures. LDT is somewhat challenging because normal (solid) foods are not allowed during the period of treatment. Both steroids and LDT are widely used - steroids predominately in the USA and LDT elsewhere. There is controversy as to which is best. This study aims to determine which should be preferred.

In this clinical study, children presenting with Crohn's disease will be randomly assigned to either steroid treatment or LDT and followed up for a period of one year. During that time the assigned treatment will be used for any episodes of active disease. We will study a total of 80 children attending the Paediatric Gastroenterology Units in Birmingham, Bristol, Liverpool, Oxford, Sheffield and St. George's Hospital in London. Various outcomes will be compared in the two groups. We will examine the recovery rates (success in bringing about remission) and the frequency of subsequent relapses. We will compare growth and physical development, because active Crohn's disease and possibly steroids may have adverse effects on these processes. A special focus of the study will be on the effect of the disease and its treatment on bone health. Using special blood and urine tests and bone scans we will compare bone growth and density in the two groups. Finally, it is crucially important that we consider the impact of the disease and its treatment on the young person on the basis of their own individual perspective. To do this we will compare the 'quality of life' of children in the two treatment groups, using a questionnaire specially designed to measure this aspect in young people with Crohn's disease.

This study will thus enable us to undertake a comprehensive comparison of the two major first-line treatments used in childhood Crohn's Disease. This is crucially important, and no such study has previously been undertaken

ELIGIBILITY:
Inclusion Criteria:

* Active Crohn's Disease with PCDAI > 20
* Aged 7 - 17 with possibility of 1 year follow-up

Exclusion Criteria:

* Previous treatment for Crohn's Disease with liquid diet or glucocorticoid therapy
* Isolated orofacial granulomatosis
* Intravenous glucocorticoid therapy immediately indicated
* Planned surgical intervention for CD

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density change based on DXA measurement at 1 year | 12 months post-recruitment

SECONDARY OUTCOMES:
Proportion in remission | 6 weeks
Change in PCDAI, HAB and pHBS | 6 weeks
Quality of life throughout treatment period, using IMPACT III measurements | 12 months
Baseline urine 11B-HSD1 and bone formation | 6 weeks
Baseline urine 11B-HSD1 activity and change in bone mineral density | 12 months
Change in urine 11B-HSD1 activity and PCDAI in patients before and after treatment with LDT and CST | 12 months
Growth impairment | 12 months
Adherence to randomised therapy for relapses | 12 months
Adverse effects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: M. Stephen Murphy, Study Director — University of Birmingham
Locations (6):
- United Kingdom (6):
  - Bristol Royal Hospital for Sick Children, Bristol, Bristol
  - St George's University Hospital, London, London
  - Royal Liverpool Children's Hospital, Liverpool, Merseyside
  - Oxford Children's Hospital, Oxford, Oxfordshire
  - Sheffield Children's Hospital, Sheffield, South Yorkshire
  - Birmingham Children's Hospital, Birmingham, West Midlands